CLINICAL TRIAL: NCT03089814
Title: Changes in Tissue Microcirculation During Ischemic Conditioning: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RIPC-VOT
Record Dates: First submitted 2017-03-14; First posted 2017-03-24 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Microcirculation
Keywords: tissue oxygen saturation, ischemic conditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Active Comparator): Healthy male volunteers will receive ischemic conditioning (4 cycles of 5-min ischemia followed by 5-min reperfusion on upper extremity) while measuring changes in tissue microcirculation at the thenar muscle.
  Interventions: Procedure: ischemic conditioning
- Cardiac surgery patients (Active Comparator): Patients scheduled for cardiac surgery will receive ischemic conditioning (4 cycles of 5-min ischemia followed by 5-min reperfusion on upper extremity) while measuring changes in tissue microcirculation at the thenar muscle.
  Interventions: Procedure: ischemic conditioning

INTERVENTIONS:
Procedure: ischemic conditioning — Four cycles of 5-min inflation of pneumatic cuff on upper extremity up to 200 mmHg, followed by 5-min deflation with no pressure.

SUMMARY:
Changes in tissue microcirculation during ischemic conditioning (4 cycles of 5-min ischemia and 5-min reperfusion) has not been well documented. In previous studies, there was difference in changes in microcirculation, such as recovery slope and occlusion slope, between healthy subjects and cardiac surgery patients. Moreover, the occlusion slope, which reflects local tissue oxygen consumption during ischemic period, is anticipated to decrease during repeated ischemia-reperfusion cycle by its protecting effect, however there has not been well-conducted study. The purpose of the study is to evaluate the changes in microcirculation measured by tissue oxygen saturation during ischemic conditioning between healthy volunteers and cardiac surgery patients.

DETAILED DESCRIPTION:
Subjects who are male healthy volunteers (aged 20-45) or who are scheduled to receive cardiac surgery (aged 20-80) will undergo ischemic conditioning, consisting of 4 cycles of 5-min ischemia with pressure of 200 mmHg on upper extremity followed by 5-min reperfusion with no pressure. During ischemic conditioning, changes in tissue microcirculation (baseline tissue saturation, occlusion slope during ischemia, and recovery slope during reperfusion) will be observed using tissue oxygen saturation sensor attached to the thenar muscle of the hand. For cardiac surgery patients, the study will be conducted before anesthesia induction on the surgery day to exclude any potential effect of anesthetics.

ELIGIBILITY:
<Healthy volunteers>

Inclusion Criteria:

* Age 20-45
* No underlying chronic disease
* Male volunteer

Exclusion Criteria:

* Under taking prescription drugs
* Taking herbal medicines within 2 weeks
* Baseline systolic blood pressure > 150 mmHg or diastolic pressure > 100 mmHg
* Body mass index < 18 kg/m^2 or > 30 kg/m^2
* Vigorous exercise, excessive alcohol, smoking or caffeine within 24 hours
* Any abnormalities on upper extremities
* Do not consent to participate

<Cardiac surgery patients>

Inclusion Criteria:

* Age 20-80
* Scheduled for cardiac surgery

Exclusion Criteria:

* Baseline systolic blood pressure > 150 mmHg or diastolic pressure > 100 mmHg
* Body mass index < 18 kg/m^2 or > 30 kg/m^2
* Uncontrolled diabetes
* Under taking beta-blockers
* Severe renal dysfunction, chronic kidney disease, on hemodialysis
* Any abnormalities on upper extremities (i.e, AV fistula on arms)
* Peripheral vascular disease, peripheral neuropathy, coagulopathy
* Vigorous exercise, excessive alcohol, smoking or caffeine within 24 hours
* Pregnant
* Emergency surgery
* Do not consent to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Changes in microcirculation during ischemic conditioning | During 4-cycles of 5-min ischemia followed by 5-min reperfusion
  Changes in occlusion slope during ischemia and recovery slope during reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No